CLINICAL TRIAL: NCT02898792
Title: Opioid Sensitivity in Adults With Treated and Untreated Obstructive Sleep Apnea
Brief Title: Remifentanil in Adults With OSA
Acronym: AROSA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201605158
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Apnea, Sleep
Keywords: sensitivity, opioid
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypersensitivity | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- targeted infusion of remifentanil untreated OSA (Experimental): Stepped-dose, targeted infusion of remifentanil with measurement of miosis, respiratory rate, end-expired CO2, and thermal analgesia and plasma drug concentrations. Remifentanil dose will be based on ideal body weight.
  Interventions: Drug: Targeted infusion of remifentanil
- targeted infusion of remifentanil CPAP treated OSA (Experimental): Stepped-dose, targeted infusion of remifentanil with measurement of miosis, respiratory rate, end-expired CO2, and thermal analgesia and plasma drug concentrations. Remifentanil dose will be based on ideal body weight.
  Interventions: Drug: Targeted infusion of remifentanil
- targeted infusion of remifentanil No OSA (Experimental): Stepped-dose, targeted infusion of remifentanil with measurement of miosis, respiratory rate, end-expired CO2, and thermal analgesia and plasma drug concentrations. Remifentanil dose will be based on ideal body weight.
  Interventions: Drug: Targeted infusion of remifentanil

INTERVENTIONS:
Drug: Targeted infusion of remifentanil — Remifentanil dosing will be calculated using ideal body weight and infused to achieve brain concentrations of 0.5, 1, 2, 3, and 4 ng/ml; approximately 10 minutes at each concentration.
  Other Names: Ultiva

SUMMARY:
Obstructive Sleep Apnea (OSA) is the most common problem that affects sleep. People with this problem have their airway blocked or minimized, causing snoring or gasping while sleeping. It can also reduce the amount of oxygen that circulates in the blood of people affected by it. Millions of Americans have OSA; 10% of adults have diagnosed OSA, an estimated 25% have undiagnosed OSA. There is concern in the medical community about how to manage pain in patients with OSA because of the risk of decreased or slower breathing associated with certain pain medications called opioids. Giving OSA patients opioids could cause them to have even lower oxygen amounts in their blood stream. It is conceivable that patients with OSA may require lower doses of opioids to cause decreased breathing as compared to patients without OSA, however this has not been proven. In this study, we are using a very short acting and easily reversible opioid pain medication called remifentanil in patients with OSA in order to find out if treated and untreated OSA patients respond to opioid differently than patients without OSA.

DETAILED DESCRIPTION:
Open-label, parallel group study. Twenty adults each with untreated OSA, CPAP-treated OSA, and no OSA will undergo a stepped-dose target-controlled opioid (remifentanil) infusion, measurement of opioid effects (miosis, respiratory rate, end-expired CO2, thermal analgesia) and plasma drug concentrations. Remifentanil clinical effects, pharmacodynamics (concentration-effect relationships), and pharmacokinetics will be compared between the three groups, as will relationships between effects and nighttime hypoxemia (assessed by home PSG).

The ultimate long-term goal for this research is to improve the perioperative care and pain management of patients with obstructive sleep apnea (OSA). While patients with OSA are believed to be more sensitive to the analgesic and adverse effects of opioids, there are no studies that assess the effects of the OSA gold-standard treatment, namely CPAP, on this purported sensitivity. Furthermore, OSA is a heterogeneous disease and not all patients who carry an OSA diagnosis are likely to have the same opioid sensitivity. At present no easily administered test is able to determine the degree of opioid sensitivity of an individual patient.

The specific goal of this research is to validate or refute, the untested yet "conventional wisdom" that adults with untreated OSA have increased sensitivity to the clinical effects of opioids, especially ventilatory depression. We will test the presumptive hypotheses that a) untreated OSA increases ventilatory, miotic, and analgesic effects of opioids, b) the magnitude of increase is proportional to the degree of nighttime hypoxia, and c) CPAP treatment of OSA normalizes altered opioid responses.

These hypotheses will be tested by evaluating the pharmacodynamics (concentration-effect relationship) of the prototype opioid remifentanil in patients with and without OSA using objective opioid sensitivity markers to determine if patients with OSA have increased sensitivity to opioids and to determine if treatment with CPAP alters this purported sensitivity. Our study drug, remifentanil, is an ultra-short acting μ-selective opioid agonist, which is the same receptor at which longer acting opioids such as morphine act. Since the site of action of remifentanil is the same as other opioids, the results of this study will be able to be generalized to other opioids, improving our clinical understanding and practice in this patient population. Opioid effects will be determined by the decrease in pupil diameter, which is the most sensitive measure of opioid effects at the drug concentrations and subanesthetic doses to be used. The degree to which changes in pupil diameter correlate with changes in respiratory rate will be compared.

ELIGIBILITY:
Inclusion Criteria

1. 18 to 70 year-old males or non-pregnant females
2. Provide informed consent

Exclusion Criteria

1. History of liver disease
2. pregnant or nursing females
3. known history of addiction to drugs or alcohol
4. craniofacial anomalies that preclude proper fit of pupillometry goggles
5. eye abnormalities that preclude the measurement of pupil diameter
6. use of home oxygen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
The relationship between remifentanil concentration and miotic effect | Baseline, 10, 20, 30, 40, and 50 minutes for each concentration

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maharaj AR, Montana MC, Hornik CP, Kharasch ED. Opioid use in treated and untreated obstructive sleep apnoea: remifentanil pharmacokinetics and pharmacodynamics in adult volunteers. Br J Anaesth. 2025 Mar;134(3):681-692. doi: 10.1016/j.bja.2024.10.042. Epub 2025 Jan 20. PMID 39837697
- [Derived] Montana MC, McLeland M, Fisher M, Juriga L, Ercole PM, Kharasch ED. Opioid sensitivity in treated and untreated obstructive sleep apnoea: a prospective cohort study. Br J Anaesth. 2024 Jan;132(1):145-153. doi: 10.1016/j.bja.2023.09.032. Epub 2023 Nov 7. PMID 37945413